CLINICAL TRIAL: NCT01844401
Title: Comparison of the Pharmacokinetic and Pharmacodynamic Profiles of Albuterol Spiromax® and ProAir® HFA in Pediatric Patients With Persistent Asthma
Brief Title: Pharmacokinetic and Pharmacodynamic Profiles of Albuterol Spiromax® and ProAir® Hydrofluoroalkane (HFA) in Pediatric Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABS-AS-102
Record Dates: First submitted 2013-04-19; First posted 2013-05-01 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Asthma
Keywords: persistent asthma; Albuterol Spiromax®; ProAir® HFA; Pediatric Patients; Phase 1
MeSH Terms: conditions — Asthma | interventions — Procaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spiromax/ProAir (Experimental): Single dose of Albuterol Spiromax® 180 mcg followed by a 4 to 14 day washout period then a single dose of ProAir® HFA 180 mcg
  Interventions: Drug: Albuterol Spiromax®; Drug: ProAir® HFA
- ProAir/Spiromax (Experimental): Single dose of ProAir® HFA 180 mcg followed by a 4 to 14 day washout period then a single dose of Albuterol Spiromax® 180 mcg
  Interventions: Drug: Albuterol Spiromax®; Drug: ProAir® HFA

INTERVENTIONS:
Drug: Albuterol Spiromax® — Albuterol Spiromax® 180 mcg (administered as 2 actuations of 90 mcg of albuterol base/actuation ex-mouthpiece) orally inhaled, single dose
  Other Names: Spiromax®
Drug: ProAir® HFA — ProAir® HFA 180 mcg (administered as 2 actuations of 90 mcg of albuterol base/actuation ex-mouthpiece) orally inhaled, single dose
  Other Names: ProAir®

SUMMARY:
The primary objective of this study is to compare the pharmacokinetic (PK) profiles of Albuterol Spiromax® and ProAir HFA after administration of a single inhaled dose of 180 mcg albuterol base from each product.

DETAILED DESCRIPTION:
This is a single center, open-label, 2-period crossover study. The study consists of a screening visit followed by a treatment period comprising 2 treatment visits. The treatment period visits will be separated by a 4 to 14-day washout period. Eligible patients will be kept overnight prior to each treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent signed and dated by the patient and/or parent/caregiver/legal guardian (as appropriate) before conducting any study-related procedure.
2. Male or pre-menarchal female patient 4-11 years of age, inclusive, as of the Screening Visit (SV)
3. Has a documented physician diagnosis of persistent asthma of a minimum of 3 months duration that has been stable for at least 4 weeks prior to the SV. The asthma diagnosis must be in accordance with the National Asthma Education and Prevention Program Guidelines Expert Panel Report 3 (EPR3).
4. Forced expiratory volume in 1 second (FEV1) >80% predicted for age, height and gender and race at the SV based on the pediatric population standards.
5. Any patient being treated with inhaled corticosteroids (ICS) must be on a lowdose regimen (200 mcg or less of fluticasone propionate per day or equivalent), which has been stable for at least 4 weeks prior to the SV and which is expected to be maintained for the duration of the study
6. Has required less than 4 inhalations per week of a rescue bronchodilator (on average) for the 4 weeks preceding the SV
7. Has the ability to withhold inhaled albuterol for at least 72 hours preceding each Treatment Visit (TV).

   * Other criteria apply, including must weigh at least 45 pounds

Exclusion Criteria:

1. A known hypersensitivity to albuterol or any of the excipients in the inhaler formulations (lactose, ethanol, etc.)
2. Participation (receiving study drug) in any investigational drug trial within the 30 days preceding the SV or planned participation in another investigational drug trial at any time during this trial
3. History of severe milk protein allergy
4. Proneness to orthostatic dysregulation, syncope, or blackouts
5. History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, acute or chronic sinusitis, otitis media, influenza) that has not resolved within 2 weeks preceding the SV.
6. History of life-threatening asthma or that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures
7. Any asthma exacerbation requiring systemic corticosteroids within 3 months of the SV. A patient must not have had any hospitalization for asthma within 6 months prior to the SV.

   * Other criteria apply.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma albuterol concentration-time curve | Time 0 to the last detectable plasma albuterol concentration measured up to 10 hours post-dose (AUC0-t)
  Blood samples for plasma albuterol concentration determination will be drawn 5 (±2) minutes prior to dosing and at 30 (±2), 60 (±5), 120 (±10), 360 (±10), and 600 (±10) minutes after the completion of dosing.
Maximum observed plasma albuterol concentration (Cmax) | From baseline to up to 10 hours post dose
  Blood samples for plasma albuterol concentration determination will be drawn 5 (±2) minutes prior to dosing and at 30 (±2), 60 (±5), 120 (±10), 360 (±10), and 600 (±10) minutes after the completion of dosing.

SECONDARY OUTCOMES:
Pharmacodynamic Effect on Vital Signs | From baseline to up to 6 hours post dose
  Effects on vital signs (blood pressure, pulse rate) over 6 hours post-dosing
Summary of participants with adverse events | From Day 1 to end of Follow-up Visit (approximately 4 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Teva Investigational Site 10538, Costa Mesa, California, United States